CLINICAL TRIAL: NCT03355898
Title: Acute Coronary Syndrome With ST Elevation in Northern Lorraine: Evolution of Clinicals, Epidemiological and Angiographic Data Since 2005
Brief Title: Acute Coronary Syndome With ST Elevation in Northern Lorraine
Acronym: StemiLor
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-06Obs-CHRMT
Record Dates: First submitted 2017-11-23; First posted 2017-11-28 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lorraine is one of the most affected French region by cardiovascular diseases with a mortality rate for ischemic heart disease higher than the national average in 2010. Due to practice change with the new recommandations of the European Society of Cardiology involving the myocardic revascularization, the investigators wanted to compare the Stemi care in 2005-2006, 2010-2011 and 2015 in the CHR Metz-Thionville.

DETAILED DESCRIPTION:
This monocentric study evaluate the impact of the new recommandations of the European Society of Cardiology in the acute coronary syndrome with ST elevation (Stemi) care. Data is compiled retrospectively from angiographic report and informatic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an acute coronary syndrome with ST elevation for less than 12 hours
* Patients with coronarography in a context of cardiorespiratory arrest with unknown cause and acute coronary occlusion

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an acute coronary syndrome with ST elevation in the CHR Metz-Thionville in 2005-2006, 2010-2011 and 2015
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Acute coronary syndrome with ST elevation care | Day 1
  Percentage of per-cutaneous angioplasty and percentage of pre-hospital thrombolysis

SECONDARY OUTCOMES:
Stenting procedure | Day 1
  Percentage of manual thrombectomy and percentage of direct stenting
Hospital mortality | Day 1
  Percentage of death during the STEMI care
Epidemiology data | Day 1
  Mean age of STEMI patients